CLINICAL TRIAL: NCT03982329
Title: Evaluation of the Benefit of Navigated Repetitive Transcranial Magnetic Stimulation for Therapy of Surgery-related Motor Deficits in Brain Tumor Patients
Brief Title: Impact of nrTMS Therapy on the Progress of Neurorehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Sandro M. Krieg, Attending Neurosurgeon, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12/15S
Record Dates: First submitted 2019-05-17; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Transcranial Magnetic Stimulation, Repetitive
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: 2/3 nrTMS, 1/3 sham
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nrTMS group (Active Comparator): 15 minutes low-frequency nrTMS (1 Hz) of the uneffected hemisphere at 7 consecutive days
  Interventions: Device: navigated repetitive transcranial magnetic stimulation; Procedure: physical therapy
- sham group (Sham Comparator): 15 minutes sham stimulation of the uneffected hemisphere at 7 consecutive days
  Interventions: Procedure: physical therapy

INTERVENTIONS:
Device: navigated repetitive transcranial magnetic stimulation
  Arms: nrTMS group
Procedure: physical therapy

SUMMARY:
Low-frequency navigated repetitive transcranial magnetic stimulation (nrTMS) of the non-damaged hemisphere to increase cortical excitability of the damaged hemisphere and to reduce the increased neuronal inhibition in patients suffering from new surgery-related paresis after brain tumor resection

DETAILED DESCRIPTION:
Postoperative loss of motor function greatly impairs the patients' quality of life and life expectancy of patients with brain tumors is significant limited. Hence the reduction of time spent on neurorehabilitation is very important.

Inclusion of patients that underwent brain tumor resection with a surgery-related paresis of the upper extremity.

Randomized controlled and double blinded trial - 2/3 nrTMS, 1/3 sham. Fifteen minutes low-frequency nrTMS (1 Hz) of the uneffected hemisphere at 7 consecutive days: nrTMS group or sham group. Thirty minutes physical therapy of the upper extremity in both groups.

MRI, nTMS motor mapping, assessments for motor status of upper extremity including Fugl-Meyer-Assessment (FMA), National Institution of Health Stroke Scale (NIHSS), Jebsen Taylor Hand Function Test (JTHFT), Nine Hole Peg Test (NHPT), and Karnofsky Performance Scale (KPS) postoperatively, after the 7th day of intervention and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* New surgery-related paresis of upper extremity after brain tumor resection
* Written informed consent for participation

Exclusion Criteria:

* Contraindications for MRI
* Contraindications for nrTMS
* Only biopsy instead of tumor resection
* Patients without preserved MEP response as measured by postoperative nTMS motor mapping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change of Fugl-Meyer Assessment (FMA) | Between first day of intervention and 3-months follow up
  Assessment upper extremity

SECONDARY OUTCOMES:
Nine Hole Peg Test (NHPT) | First day of intervention = postoperatively, after the 7th day of intervention and after 3 months
  Fine motor skills upper extremity
National Institutes of Health Stroke Scale (NIHSS) | First day of intervention = postoperatively, after the 7th day of intervention and after 3 months
  The scale measures neurological outcome; Total score is reported; Scores on the NIHSS range from 0 to 42, with higher scores indicating more severe disability
Jebsen Taylor Hand Function Test (JTHFT) | First day of intervention = postoperatively, after the 7th day of intervention and after 3 months
  Functionality upper extremity
Karnofsky Performance Status (KPS) | First day of intervention = postoperatively, after the 7th day of intervention and after 3 months
  The scale measures general oncological outcome; the total score is reported; Scores on the KPS scale range from 0% to 100%, with higher scores indicating less disability and and better quality of life in cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Sandro M. Krieg, MD, Principal Investigator — Department of Neurosurgery, School of Medicine, TU Munich
Locations (1):
- Department of Neurosurgery, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ille S, Kelm A, Schroeder A, Albers LE, Negwer C, Butenschoen VM, Sollmann N, Picht T, Vajkoczy P, Meyer B, Krieg SM. Navigated repetitive transcranial magnetic stimulation improves the outcome of postsurgical paresis in glioma patients - A randomized, double-blinded trial. Brain Stimul. 2021 Jul-Aug;14(4):780-787. doi: 10.1016/j.brs.2021.04.026. Epub 2021 May 11. PMID 33984536